CLINICAL TRIAL: NCT04387318
Title: Effects of Inspiratory Muscle Training and Neuromuscular Electrical Stimulation in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Inspiratory Muscle Training and Neuromuscular Electrical Stimulation in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Isabella Martins de Albuquerque, Principal Investigator, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08527219.0.0000.5346
Record Dates: First submitted 2020-05-01; First posted 2020-05-13 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Multimodal training (Experimental): IMT + NMES + Pulmonary Rehabilitation
  IMT will be performed using a device with linear load pressure (POWERbreathe Medic Plus ®, SP, BR).
  NMES will be applied using an calibrated electrical stimulator (Neurodyn High Volt, IBRAMED, São Paulo/São Paulo, Brazil).
  Pulmonary Rehabilitation: The physical training part of pulmonary rehabilitation will consist of aerobic and resistance exercise.
  Interventions: Device: Multimodal training
- IMT + Pulmonary Rehabilitation (Experimental): IMT will be performed using a device with linear load pressure (POWERbreathe Medic Plus ®, SP, BR).
  Pulmonary Rehabilitation: The physical training part of pulmonary rehabilitation will consist of aerobic and resistance exercise.
  Interventions: Device: IMT + Pulmonary Rehabilitation
- NMES + Pulmonary Rehabilitation (Experimental): NMES will be applied using an calibrated electrical stimulator (Neurodyn High Volt, IBRAMED, São Paulo/São Paulo, Brazil).
  Pulmonary Rehabilitation: The physical training part of pulmonary rehabilitation will consist of aerobic and resistance exercise.
  Interventions: Device: NMES + Pulmonary Rehabilitation
- Pulmonary Rehabilitation (Placebo Comparator): Pulmonary Rehabilitation: The physical training part of pulmonary rehabilitation will consist of aerobic and resistance exercise.
  Interventions: Device: Pulmonary Rehabilitation

INTERVENTIONS:
Device: Multimodal training — IMT will be performed using the POWERbreathe® Medic Plus inspiratory training device for five sets of 10 repetitions each, with a one-minute interval between each set. The initial load set will be 30% of maximal inspiratory pressure (MIP), during the first two weeks to allow for an adjustment period. The IMT wil be performed two times per week for 8 weeks.
  NMES will be applied using an calibrated electrical stimulator (Neurodyn High Volt, IBRAMED, São Paulo/São Paulo, Brazil). The following parameters will be used: 50 Hz frequency, pulse duration of 400 µs, work cycle of 5 seconds ON and 15 seconds OFF (first month) adjusted for 10 seconds ON and 30 seconds OFF (second month) and maximum intensity tolerated during 2 times per week for 8 weeks.
  Pulmonary Rehabilitation The pulmonary rehabilitation will consist of aerobic and resistance exercise during 8 weeks.
  Arms: Multimodal training
Device: IMT + Pulmonary Rehabilitation — IMT will be performed using the POWERbreathe® Medic Plus (POWERbreathe Medic Plus ®, SP, BR) inspiratory training device for five sets of 10 repetitions each, with a one-minute interval between each set. The initial load set will be 30% of maximal inspiratory pressure (MIP), during the first two weeks to allow for an adjustment period. After that, load increases occurred as follows: 35% of MIP in week 3, 40% of MIP in week 4, 45% of MIP in week 5, 50% of MIP at week 6, 55% of MIP in week 7, and 60% of MIP in weeks 8.
  Pulmonary Rehabilitation The pulmonary rehabilitation will consist of aerobic and resistance exercise during 8 weeks.
  Arms: IMT + Pulmonary Rehabilitation
Device: NMES + Pulmonary Rehabilitation — NMES will be applied using an calibrated electrical stimulator (Neurodyn High Volt, IBRAMED, São Paulo/São Paulo, Brazil). The following parameters will be used: 50 Hz frequency, pulse duration of 400 µs, work cycle of 5 seconds ON and 15 seconds OFF (first month) adjusted for 10 seconds ON and 30 seconds OFF (second month) and maximum intensity tolerated during 2 times per week for 8 weeks.
  Pulmonary Rehabilitation The pulmonary rehabilitation will consist of aerobic and resistance exercise during 8 weeks.
  Arms: NMES + Pulmonary Rehabilitation
Device: Pulmonary Rehabilitation — Pulmonary Rehabilitation The pulmonary rehabilitation will consist of aerobic and resistance exercise during 8 weeks.
  Arms: Pulmonary Rehabilitation

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a significant current public health problem, characterized by the presence of limited airflow. However, COPD has important manifestations beyond the lungs, the so-called systemic effects. These included dysfunction of peripheral and respiratory muscles. The growing amount of evidence has shown that patients with COPD also present important deficits in postural balance and consequently, increased risk of falling. As an essential part of the management of COPD, pulmonary rehabilitation (PR) alleviates dyspnea and fatigue, improves exercise tolerance and health-related quality of life, and reduces hospital admissions and mortality for COPD patients. Exercise is the key component of PR, which is composed of exercise assessment and training therapy. Currently, two modalities of therapy have been suggested as complementary to pulmonary rehabilitation: inspiratory muscular training (IMT) and neuromuscular electrical stimulation (NMES). Based on the premise that peripheral and respiratory muscle dysfunction can negatively impact postural control of patients with COPD, and given the importance of balance as a modifiable risk factor for falls, it is important to investigate whether the use of these therapeutic modalities (IMT and/or NMES) is capable of improving the short-term effects of pulmonary rehabilitation and also promoting improved balance.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD, in stages II, III and IV, according to criteria of the Global Initiative for COPD (GOLD);
* Clinically stable, i.e., absence of infections or exacerbations in the last 3 months;
* Medical team allows patient to exercise
* Availability of attending the rehabilitation program.

Exclusion Criteria:

* Unstable primary pathologies (cardiovascular, renal, metabolic, psychiatric);
* Hemodynamic instability;
* Nutritional supplementation on the 4 weeks preceding the study;
* Severe hearing or visual impairment recorded on patient chart or self-referred;
* Obesity (BMI > 30 kg/m2);
* Neurological or musculoskeletal condition that severely limits mobility and postural control, thus making it impossible to carry out the assessments;
* Electronic devices, such as heart pacemakers and implantable cardioverter defibrillator;
* Skin injuries and infection where electrodes would be placed;
* Prior participation in pulmonary rehabilitation programs 3 months previous to the study;
* Vertigo;
* Active smoker and/or alcoholic;
* Neurological impairment or cerebellar lesions;
* Deficit in cognitive function;
* Severe vitamin D deficiency;
* Physically active.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Static postural balance | Post-intervention (change after 8 weeks of training)
  Static postural balance will be assessed on a portable force platform (AccuSway Plus, AMTI®, MA, USA) using the center of pressure displacement amplitude in the anteroposterior direction (COP) (cm).
Static postural balance | Post-intervention (change after 8 weeks of training)
  Static postural balance will be assessed on a portable force platform (AccuSway Plus, AMTI®, MA, USA) using the area of ellipse (AE) (cm2).
Static postural balance | Post-intervention (change after 8 weeks of training)
  Static postural balance will be assessed on a portable force platform (AccuSway Plus, AMTI®, MA, USA) using the velocity of displacement of center of pressure (COPvel) (cm/s).
Static postural balance | Post-intervention (change after 8 weeks of training)
  Static postural balance will be assessed on a portable force platform (AccuSway Plus, AMTI®, MA, USA) using the center of area of pressure and area of ellipse (AE) (cm2).

SECONDARY OUTCOMES:
Static postural balance | Post-intervention (change after 8 weeks of training)
  Static postural balance (%) will assessed through Foam-Laser dynamic posturography.
Static and dynamic postural balance | Post-intervention (change after 8 weeks of training)
  Static and dynamic postural balance will assessed using the Berg Balance Scale (score points). Scores range from 0 to 56, with higher scores indicating better balance.
Static and dynamic postural balance | Post-intervention (change after 8 weeks of training)
  Static and dynamic postural balance will assessed using the Balance Evaluation Systems Test (score points). The total score of the test (108 points) will be calculated with a percentage score (0-100%) and higher scores indicate better balance performance.
Dynamic postural balance | Post-intervention (change after 8 weeks of training)
  Dynamic postural balance will assessed using the Timed Up and Go (seconds). A faster time indicate a better functional performance and a score of ≥12 seconds used as a cut-point.
Balance confidence questionnaire | Post-intervention (change after 8 weeks of training)
  Balance confidence questionnaire will measured through the Activities Specific Balance Confidence Scale (total score points). The questionnaire contains 16 items scored on a range from 0% to 100% (0 indicating no confidence and 100 indicating full confidence).
Balance confidence questionnaire | Post-intervention (change after 8 weeks of training)
  Balance confidence questionnaire will measured through Falls Efficacy Scale-International (total score points). The total score ranges from 16 to 64 points. Higher values indicate less fall-related self-efficacy (and more concern about falling).
Peripheral muscle strength | Post-intervention (change after 8 weeks of training)
  Handgrip strength and quadriceps muscle strength will be assessed by dynamometry, respectively, Kgf and Newtons.
Respiratory muscle strength and inspiratory muscle endurance | Post-intervention (change after 8 weeks of training)
  Respiratory muscle strength (cmH2O) and inspiratory muscle endurance (cmH2O) will measured through digital pressure manometry and incremental and constant test, respectively
Quadriceps femoris and diaphragm thickness | Post-intervention (change after 8 weeks of training)
  Quadriceps femoris and diaphragm thickness will measured by ultrasonography
Submaximal level of functional capacity | Post-intervention (change after 8 weeks of training)
  Submaximal level of functional capacity will measured by 6-minute walk test
Health-related quality of life at 8 week | Post-intervention (change after 8 weeks of training)
  Health-related quality of life will measured by Saint George's Respiratory Questionnaire. Overall scores range from 0 (no effect on quality of life) to a maximum score of 100 (maximum perceived distress).
Oxidant profile | Post-intervention (change after 8 weeks of training)
  The oxidant profile will be assessed by Dichlorofluorescein Diacetate - DCF-DA (picomoles / mL).
Oxidant profile | Post-intervention (change after 8 weeks of training)
  The oxidant profile will be assessed by Thiobarbituric Acid Reactive Substances -TBARS (nmol de MDA/mL).
Oxidant profile | Post-intervention (change after 8 weeks of training)
  The oxidant profile will be assessed by Advanced Oxidation Protein Products - AOPPs (µmol/L).
Oxidant profile | Post-intervention (change after 8 weeks of training)
  The oxidant profile will be assessed by Total Oxidant Status - TOS (mmol Trolox Equiv/L).
Antioxidant profile | Post-intervention (change after 8 weeks of training)
  The antioxidant profile will be assessed by Ferric Reducing Antioxidant Power - FRAP- (µmol/L)
Antioxidant profile | Post-intervention (change after 8 weeks of training)
  The antioxidant profile will be assessed by Total Antioxidant Capacity- CAT (mmol Trolox Equiv/L).
Muscle damage | Post-intervention (change after 8 weeks of training)
  Muscle damage will assessed through creatine phosphokinase (total CPK) (U/L).
Muscle damage | Post-intervention (change after 8 weeks of training)
  Muscle damage will assessed through lactate dehydrogenase (LDH) (U/L).
Muscle damage | Post-intervention (change after 8 weeks of training)
  Muscle damage will assessed through lactate parameter (mg/dL).
DNA damage | Post-intervention (change after 8 weeks of training)
  DNA damage will assessed by means of the Comet and micronucleus assay
Endothelial function | Post-intervention (change after 8 weeks of training)
  Endothelial function will assessed through nitrite/nitrate oxide (NOx) (µmol/L)
Peripheral muscle resistance of the lower limbs | Post-intervention (change after 8 weeks of training)
  Peripheral muscle resistance of the lower limbs will assessed through 30-second Sit-to-Stand tests (repetitions)

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Albuquerque, DSc, Study Chair — Universidade Federal de Santa Maria; Tamires dos Santos, MSc, Principal Investigator — Universidade Federal de Santa Maria; Aron Silveira, DSc, Study Chair — Universidade Federal de Santa Maria
Locations (1):
- Universidade Federal de Santa Maria, Santa Maria, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Daros Dos Santos T, Pasqualoto AS, Cardoso DM, Da Cruz IBM, Moresco RN, Ferreira da Silveira A, Martins de Albuquerque I. Effects of multimodal exercise program on postural balance in patients with chronic obstructive pulmonary disease: study protocol for a randomized controlled trial. Trials. 2023 Aug 15;24(1):532. doi: 10.1186/s13063-023-07558-9. PMID 37580800